CLINICAL TRIAL: NCT05532670
Title: SpO2 Accuracy Validation of N600x Sensors Via Reference CO-Oximetry in Healthy, Well-Perfused Subjects
Brief Title: N600X Low Saturation Accuracy Validation
Status: Completed | Type: Observational
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Other Study IDs: MDT22013LSOXMN
Record Dates: First submitted 2022-08-31; First posted 2022-09-08 (Actual); Last update posted 2022-11-23 (Actual); Status verified 2022-11

CONDITIONS: Hypoxia
Keywords: Oxygen Saturation; Invasive Controlled Desaturation; Pulse Oximetry; Desaturation of Blood
MeSH Terms: conditions — Hypoxia | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: Non-Invasive Controlled Hypoxia — Following arterial cannulation, hypoxia is induced by reducing the percent of inspired oxygen the subject breathes while simultaneous measurements are recorded from the test pulse oximeters and arterial blood samples are collected at targeted levels of saturation.
  Other Names: Desaturation; Blood Sampling

SUMMARY:
To compare pulse oximetry saturation measurements, during normal to low saturation, to saturation measurements made by a multi-wavelength CO-oximeter, taken from arterial blood samples from healthy human subjects.

DETAILED DESCRIPTION:
The study utilizes a single-site, physiology laboratory (Clinimark) to conduct this Post Market, non-randomized, prospective studies. The goal is to enroll a minimum of fifteen subjects. Subject pool goal of diversity across ethnicity, race and sex of varying skin tones to meet the study design requirements.

The general purpose of Invasive Controlled Desaturation Studies is to support the SpO2 accuracy of the post market pulse oximetry sensors and paired monitor in comparison to reference-standard measurements of blood SaO2 by a CO-oximeter during low saturation conditions. This is achieved through paired observations of SpO2 and SaO2 values over the specified SpO2 accuracy range of 60% to 100% SaO2 of the pulse oximeter on a group of healthy adult volunteers. The fraction of inspired oxygen (FiO2) delivered to test subjects is varied to achieve a series of targeted steady-state saturation periods. Arterial blood samples are periodically taken from an indwelling arterial catheter for use in the comparison. Pulse rate accuracy will be evaluated during the same data collection period as SpO2. Pulse rate will be compared to reference ECG heart rate.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must have the ability to understand and provide written informed consent

2 Adult subjects 18 to 50 years of age.

3. Subject must be willing and able to comply with study procedures and duration.

4. Subject is a non-smoker or who has not smoked within 2 days prior to the study.

5. Any gender of any race.

6. Cleared same day Health Assessment form and health screening.

7. Cleared physical exam by a licensed physician, physician assistant, or advanced practice nurse (medical exam includes 12-lead ECG, medical history and blood test to show no sickle cell disease present)

8. Successful Perfusion Index Ulnar/Ulnar+Radial Ratio test showing adequate collateral blood flow.

Exclusion Criteria:

1. Subject with sickle cell disease.
2. Subject is considered as being morbidly obese (defined as BMI >39.5)
3. Compromised circulation, injury, or physical malformation of fingers, hands, ears or forehead/skull or other sensor sites which would limit the ability to test sites needed for the study. (Note: Certain malformations may still allow subjects to participate if the condition is noted and would not affect the sites utilized.)
4. Females of childbearing potential, who are pregnant, who are trying to get pregnant or who have a urine test positive for pregnancy on the day of the study
5. Subjects with COHb levels >3% as assessed by CO-Oximetry during the procedure
6. tHb < 10 g/dl as assessed by CO-Oximetry during the procedure
7. MetHb ≥ 2% as assessed by CO-Oximetry during the procedure
8. Subjects with known respiratory conditions such as:

   1. uncontrolled / severe asthma,
   2. flu or influenza type infection
   3. pneumonia / bronchitis,
   4. shortness of breath / respiratory distress,
   5. unresolved respiratory or lung surgery,
   6. emphysema, COPD, lung disease
9. Subjects with known heart or cardiovascular conditions such as:

   1. Hypertension: systolic >140mmHg, or Diastolic >90mmHg on 3 consecutive readings.
   2. have had cardiovascular surgery
   3. Chest pain (angina)
   4. heart rhythms other than a normal sinus rhythm or respiratory sinus arrhythmia
   5. previous heart attack
   6. blocked artery
   7. unexplained shortness of breath
   8. congestive heart failure (CHF)
   9. history of stroke
   10. transient ischemic attack
   11. carotid artery disease
   12. myocardial ischemia
   13. myocardial infarction
   14. cardiomyopathy

Self-reported health conditions as identified in the Health Assessment Form

1. diabetes,
2. uncontrolled thyroid disease,
3. kidney disease / chronic renal impairment,
4. history of seizures (except childhood febrile seizures),
5. epilepsy,
6. history of unexplained syncope,
7. recent history of frequent migraine headaches,
8. recent symptomatic head injury, within the last 2 months
9. Subjects with known clotting disorders
10. history of bleeding disorders or personal history of prolonged bleeding from injury
11. history of blood clots
12. hemophilia
13. current use of blood thinner: prescription or daily use of aspirin
14. Subjects with Severe contact allergies to standard adhesives, latex or other materials found in pulse oximetry sensors, ECG electrodes, respiration monitor electrodes or other medical sensors
15. Subjects with prior or known severe allergies to lidocaine (or similar pharmacological agents, e.g. Novocain) or heparin
16. Arterial cannulation within the last 30 days prior to study date, (this may exclude only one radial artery site. Left or right)
17. History of clinically significant complications from previous arterial cannulation.
18. A radial artery with ten or more arterial cannulations right or left, excludes that site.
19. Unwillingness or inability to remove colored nail polish or colored artificial nails other than clear from test digits.
20. Other known health condition, should be considered upon disclosure in Health Assessment form

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Study Population
  The study population includes a 15 healthy non-smoking competent adults 18-50 years of age. With an aim of diversity across ethnicity, race and sex of varying skin tones.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2022-09-29 (Actual); Primary Completion 2022-10-07 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
Comparison of pulse rate (BPM) by a pulse oximeter monitor and sensor, compared to ECG pulse rate measurement | October 2022
  To validate the proposed claims for pulse rate (BPM) accuracy in diverse subject population during Low Saturation over a specified saturation ranges.
Comparison of SPO2 saturation levels by a pulse oximeter to saturation measurements made by a multi-wavelength CO-oximeter. | October 2022
  To validate the proposed claims for SPO2 saturation accuracy in diverse subject population during Low Saturation over a specified saturation ranges.

CONTACTS AND LOCATIONS:
Overall Officials: Arthur Cabrera, MD, Principal Investigator — Clinimark, LLC
Locations (1):
- Clinimark, Louisville, Colorado, United States

IPD SHARING:
Plan to Share IPD: No
All participant data will be analyzed and outlined in final study report. Individual participant data will only be made available to the participant and or participant primary care physician as applicable.